CLINICAL TRIAL: NCT00810693
Title: Randomized, Double-blind, Placebo-controlled, Multi-centre, Multi-national Study to Evaluate the Efficacy and Safety of Oral BAY63-2521 (1 mg, 1.5 mg, 2 mg, or 2.5 mg Tid) in Patients With Symptomatic Pulmonary Arterial Hypertension (PAH)
Brief Title: A Study to Evaluate Efficacy and Safety of Oral BAY63-2521 in Patients With Pulmonary Arterial Hypertension (PAH)
Acronym: PATENT-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12934; 2008-003482-68 (EudraCT Number)
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Results first posted 2014-02-26 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary arterial hypertension; PH; Stimulator
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — riociguat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT (Experimental): Participants received Riociguat orally as a film-coated tablet up to 2.5mg three times daily (tid) (titration between 1.0 mg and 2.5 mg tid based on an individual dose titration (IDT) scheme) for 12 weeks
  Interventions: Drug: Riociguat (Adempas, BAY63-2521)
- Riociguat (Adempas, BAY63-2521) up to 1.5 mg_IDT (Experimental): Participants received Riociguat orally as a film-coated tablet up to 1.5mg three times daily (tid) (titration between 1.0 mg and 1.5 mg tid based on an individual dose titration (IDT) scheme) for 12 weeks
  Interventions: Drug: Riociguat (Adempas, BAY63-2521)
- Placebo (Placebo Comparator): Participants received Placebo orally as a film-coated tablet three times daily (tid) for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riociguat (Adempas, BAY63-2521) — BAY63-2521: 1mg tid - 2.5mg tid orally for 12 weeks
  Arms: Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT
Drug: Riociguat (Adempas, BAY63-2521) — BAY63-2521: 1.5mg tid orally for 12 weeks
  Arms: Riociguat (Adempas, BAY63-2521) up to 1.5 mg_IDT
Drug: Placebo — Matching Placebo tid orally for 12 weeks
  Arms: Placebo

SUMMARY:
The aim of the study is to assess the efficacy and safety of different doses of BAY63-2521 given orally for 12 weeks, in patients with symptomatic Pulmonary Arterial Hypertension (PAH).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with symptomatic PAH (Idiopathic, Familial, Associated PAH due to connective tissue disease, congenital heart disease, portal hypertension with liver cirrhosis, or due to anorexigen or amphetamine use)
* Treatment naive patients and patients pre-treated with an Endothelin Antagonist or a Prostacyclinanalogue (except I.V.).

Exclusion Criteria:

* All types of pulmonary hypertension except subtypes of Venice Group I specified in the inclusion criteria, severe COPD (chronic obstructive pulmonary disease), uncontrolled arterial hypertension, left heart failure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2008-12-17 (Actual); Primary Completion 2012-05-14 (Actual); Study Completion 2012-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (110):
- United States (17):
  - Tucson, Arizona
  - La Jolla, California
  - Los Angeles, California
  - Sacramento, California
  - Aurora, Colorado
  - Louisville, Kentucky
  - Boston, Massachusetts
  - Omaha, Nebraska
  - New York, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Fairfield, Ohio
  - Providence, Rhode Island
  - Dallas, Texas
  - El Paso, Texas
  - Houston, Texas
- Capital Federal, Argentina
- Australia (6):
  - Darlinghurst, New South Wales
  - New Lambton Heights, New South Wales
  - Auchenflower, Queensland
  - Herston, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Prahran, Victoria
- Austria (3):
  - Linz, Upper Austria
  - Innsbruck
  - Vienna
- Belgium (2):
  - Bruxelles - Brussel
  - Leuven
- Brazil (3):
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
  - Rio de Janeiro
- Canada (3):
  - Calgary, Alberta
  - Toronto, Ontario
  - Montreal, Quebec
- China (3):
  - Guangzhou, Guangdong
  - Beijing
  - Shanghai
- Prague, Czechia
- Aarhus N, Denmark
- France (8):
  - Besançon
  - Brest
  - Grenoble
  - Lille
  - Montpellier
  - Nice
  - Pessac
  - Rouen
- Germany (9):
  - Heidelberg, Baden-Wurttemberg
  - München, Bavaria
  - Giessen, Hesse
  - Hanover, Lower Saxony
  - Greifswald, Mecklenburg-Vorpommern
  - Cologne, North Rhine-Westphalia
  - Homburg, Saarland
  - Dresden, Saxony
  - Leipzig, Saxony
- Chaïdári, Greece
- Petah Tikva, Israel
- Italy (5):
  - Trieste, Friuli Venezia Giulia
  - Rome, Lazio
  - Milan, Lombardy
  - Pavia, Lombardy
  - Turin, Piedmont
- Japan (15):
  - Nagoya, Aichi-ken
  - Yoshida, Fukui
  - Kobe, Hyōgo
  - Toride, Ibaraki
  - Tsukuba, Ibaraki
  - Kanazawa, Ishikawa-ken
  - Sagamihara, Kanagawa
  - Sendai, Miyagi
  - Tomigusuku, Okinawa
  - Bunkyo-ku, Tokyo
  - Mitaka, Tokyo
  - Ōta-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Hiroshima
  - Okayama
- Mexico (5):
  - Guadalajara, Jalisco
  - Monterrey, Nuevo León
  - Culiacán, Sinaloa
  - Mexico City
  - Querétaro
- Christchurch, New Zealand
- Otwock, Poland
- Portugal (3):
  - Coimbra
  - Lisbon
  - Porto
- Russia (2):
  - Moscow
  - Saint Petersburg
- Singapore, Singapore
- South Korea (2):
  - Seoul, Seoul Teugbyeolsi
  - Seoul
- Spain (2):
  - Barcelona
  - Seville
- Sweden (3):
  - Linköping
  - Lund
  - Umeå
- Zurich, Switzerland
- Taiwan (2):
  - Kaohsiung City
  - Taipei
- Thailand (2):
  - Bangkok
  - Chiang Mai
- Turkey (Türkiye) (3):
  - Ankara
  - Istanbul
  - Izmir
- United Kingdom (3):
  - Cambridge, Cambridgeshire
  - Clydebank, West Dunbartonshire
  - London

REFERENCES:
- [Result] Archer SL. Riociguat for pulmonary hypertension--a glass half full. N Engl J Med. 2013 Jul 25;369(4):386-8. doi: 10.1056/NEJMe1306684. No abstract available. PMID 23883383
- [Result] Ghofrani HA, Galie N, Grimminger F, Grunig E, Humbert M, Jing ZC, Keogh AM, Langleben D, Kilama MO, Fritsch A, Neuser D, Rubin LJ; PATENT-1 Study Group. Riociguat for the treatment of pulmonary arterial hypertension. N Engl J Med. 2013 Jul 25;369(4):330-40. doi: 10.1056/NEJMoa1209655. PMID 23883378
- [Result] Rosenkranz S, Ghofrani HA, Beghetti M, Ivy D, Frey R, Fritsch A, Weimann G, Saleh S, Apitz C. Riociguat for pulmonary arterial hypertension associated with congenital heart disease. Heart. 2015 Nov;101(22):1792-9. doi: 10.1136/heartjnl-2015-307832. Epub 2015 Jul 1. PMID 26135803
- [Result] Wang C, Jing ZC, Huang YG, Zhou DX, Liu ZH, Meier C, Nikkho S, Curram J, Zhang P, He JG. Riociguat for the treatment of pulmonary hypertension: Chinese subgroup analyses and comparison. Heart Asia. 2016 May 17;8(1):74-82. doi: 10.1136/heartasia-2015-010712. eCollection 2016. PMID 27326239
- [Result] Ghofrani HA, Humbert M, Langleben D, Schermuly R, Stasch JP, Wilkins MR, Klinger JR. Riociguat: Mode of Action and Clinical Development in Pulmonary Hypertension. Chest. 2017 Feb;151(2):468-480. doi: 10.1016/j.chest.2016.05.024. Epub 2016 Jun 2. PMID 27263466
- [Result] Benza RL, Boucly A, Farber HW, Frost AE, Ghofrani HA, Hoeper MM, Lambelet M, Rahner C, Bansilal S, Nikkho S, Meier C, Sitbon O. Change in REVEAL Lite 2 risk score predicts outcomes in patients with pulmonary arterial hypertension in the PATENT study. J Heart Lung Transplant. 2022 Mar;41(3):411-420. doi: 10.1016/j.healun.2021.10.013. Epub 2021 Oct 28. PMID 34848133
- [Result] Benza RL, Farber HW, Frost AE, Ghofrani HA, Corris PA, Lambelet M, Nikkho S, Meier C, Hoeper MM. Application of the REVEAL risk score calculator 2.0 in the CHEST study. Respir Med. 2022 Apr-May;195:106783. doi: 10.1016/j.rmed.2022.106783. Epub 2022 Mar 1. PMID 35256218
- [Derived] Benza RL, Ghofrani HA, Grunig E, Hoeper MM, Jansa P, Jing ZC, Kim NH, Langleben D, Simonneau G, Wang C, Busse D, Meier C, Ghio S. Effect of riociguat on right ventricular function in patients with pulmonary arterial hypertension and chronic thromboembolic pulmonary hypertension. J Heart Lung Transplant. 2021 Oct;40(10):1172-1180. doi: 10.1016/j.healun.2021.06.020. Epub 2021 Jul 10. PMID 34353714
- [Derived] Humbert M, Coghlan JG, Ghofrani HA, Grimminger F, He JG, Riemekasten G, Vizza CD, Boeckenhoff A, Meier C, de Oliveira Pena J, Denton CP. Riociguat for the treatment of pulmonary arterial hypertension associated with connective tissue disease: results from PATENT-1 and PATENT-2. Ann Rheum Dis. 2017 Feb;76(2):422-426. doi: 10.1136/annrheumdis-2015-209087. Epub 2016 Jul 25. PMID 27457511
- [Derived] Saleh S, Becker C, Frey R, Muck W. Population pharmacokinetics and the pharmacokinetic/pharmacodynamic relationship of riociguat in patients with pulmonary arterial hypertension or chronic thromboembolic pulmonary hypertension. Pulm Circ. 2016 Mar;6(Suppl 1):S86-96. doi: 10.1086/685404. PMID 27162632
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/12934

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only participants with symptomatic Pulmonary arterial hypertension (PAH) could participate in this study. Both treatment-naïve participants and participants pre-treated with an endothelin receptor antagonist or a non-intravenous prostacyclin analogue could be included.
Pre-assignment Details: 586 participants were enrolled in 124 study centers in 30 countries worldwide. 141 of the 586 enrolled participants were not randomized (adverse event [4], protocol violation [129], withdrawal by subject [8]). 445 of the 586 participants were randomized. 443 of the 445 randomized participants received study medication.
Period: Treatment Period
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Riociguat (Adempas, BAY63-2521) up to 1.5 mg_IDT | Placebo
Started | 254 | 64 (1 randomized but not treated) | 127 (1 randomized but not treated)
Participants Received Treatment | 254 | 63 | 126
Completed | 237 | 57 | 111
Not Completed | 17 | 7 | 16
Not completed — Adverse Event | 8 | 1 | 7
Not completed — Death | 0 | 1 | 2
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Non-compliance | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 2
Not completed — Withdrawal by Subject | 6 | 2 | 3
Not completed — Not treated | 0 | 1 | 1
Period: Follow-up Period (FUP)
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Riociguat (Adempas, BAY63-2521) up to 1.5 mg_IDT | Placebo
Started | 23 (Started FUP only if prematurely withdrawn from trt period or if not entering LTE study.) | 7 (Started FUP only if prematurely withdrawn from trt period or if not entering LTE study.) | 16 (Started FUP only if prematurely withdrawn from trt period or if not entering LTE study.)
Completed | 15 | 4 | 12
Not Completed | 8 | 3 | 4
Not completed — Adverse Event | 3 | 1 | 1
Not completed — Death | 2 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Riociguat (Adempas, BAY63-2521) up to 1.5 mg_IDT | Placebo | Total
Number analyzed (Participants) | 254 | 63 | 126 | 443
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.1 (16.6) | 48.8 (16.1) | 50.7 (16.5) | 50.6 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 203 | 49 | 98 | 350
  Male | 51 | 14 | 28 | 93
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 161 | 33 | 78 | 272
  Black or African American | 4 | 1 | 1 | 6
  Asian | 79 | 22 | 38 | 139
  Mixed | 1 | 0 | 1 | 2
  Not reported | 9 | 7 | 8 | 24
Prior PH therapy [Number; unit: Participants]
  Therapy-Naive | 123 | 32 | 66 | 221
  Pre-Treated | 131 | 31 | 60 | 222
pre-treated with endothelin receptor antagonist [Number; unit: Participants] — Subjects pre-treated with an endothelin receptor antagonist.
  Participants
    Yes | 113 | 27 | 54 | 194
    No | 141 | 36 | 72 | 249
pre-treated with prostacyclin analogue [Number; unit: Participants] — Subjects pre-treated with a prostacyclin analogue.
  Participants
    Yes | 20 | 4 | 7 | 31
    No | 234 | 59 | 119 | 412
PAH subtype [Number; unit: Participants] — Subtypes acc. to the Venice Clinical Classification of PH, Group 1 (idiopathic PAH, familial PAH, associated PAH due to [1] connective tissue disease, [2] congenital heart disease, [3] portal hypertension with liver cirrhosis, or [4] anorexigen or amphetamine use)
  Participants
    Idiopathic PAH | 149 | 39 | 84 | 272
    Familial PAH | 7 | 1 | 1 | 9
    Connective tissue disease assoc. PAH | 71 | 15 | 25 | 111
    Congenital heart disease (operated) assoc. PAH | 15 | 8 | 12 | 35
    Portal Pulmonary hypertension | 11 | 0 | 2 | 13
    Anorexigen or Amphtamin assoc: PAH | 1 | 0 | 2 | 3
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.91 (5.48) | 26.85 (5.35) | 26.26 (5.92) | 26.14 (5.59)
Baseline 6MWD [Mean (Standard Deviation); unit: meters] — 6-minute walking distance (6MWD) is a measure for the objective evaluation of a patient's functional exercise capacity.
  meters | 361.4 (67.7) | 363.2 (66.6) | 367.8 (74.6) | 363.5 (69.5)
WHO (World Health Organization) functional class [Number; unit: Participants] — The WHO functional assessment of pulmonary arterial hypertension ranged from functional class I (participants with PH but without resulting limitation of physical activity) to class IV (participants with PH with inability to carry out any physical activity without symptoms. These participants manifest signs of right-heart failure.). Changes to a lower WHO functional class resemble improvement; changes to a higher functional class resemble deterioration of PAH.
  Participants
    I | 5 | 5 | 4 | 14
    II | 108 | 19 | 60 | 187
    III | 140 | 39 | 58 | 237
    IV | 1 | 0 | 3 | 4
    missing | 0 | 0 | 1 | 1
Pulmonary vascular resistance [Mean (Standard Deviation); unit: dn*s*cm^-5] — The pulmonary vascular resistance (PVR) is a calculated hemodynamic parameter. PVR is derived from the directly measured parameters mean pulmonary arterial pressure (PAPmean) and pulmonary capillary wedge pressure (PCWP), divided by the cardiac output (CO). PVR and PAPmean are acquired during a right heart catheterization. CO is a calculated hemodynamic parameter, too. Formula: PVR = 80*(PAPmean - PCWP)/CO
  dn*s*cm^-5 | 790.96 (452.60) | 847.81 (548.17) | 834.06 (476.71) | 810.89 (473.45)

OUTCOME MEASURES:

1. Primary Outcome: 6 Minutes Walking Distance (6MWD) - Change From Baseline to Week 12
Description: 6-minute walking distance (6MWD) is a measure for the objective evaluation of a patient's functional exercise capacity.
Time Frame: Baseline and week 12
Population: Intent to Treat (ITT) - a randomized participant was valid for ITT analyses if at least one dose of study medication was administered.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Riociguat (Adempas, BAY63-2521) up to 1.5 mg_IDT | Placebo
Number analyzed (Participants) | 254 | 63 | 126
Meters | 29.6 (65.8) | 31.1 (79.3) | -5.6 (85.5)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT vs Placebo; Missing values for participants who withdrew/died before 12 weeks were imputed with worst value of 0m in case of death or clinical worsening without termination visit and with last observed value otherwise. Comparison was done using ANCOVA, with baseline 6MWD as a covariate and treatment group, region and treatment naive/add-on therapy as main effects. The primary statistical method was the stratified Wilcoxon test if the Shapiro-Wilk test for normality of residuals was statistically significant; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Prespecified significance level for all significance tests was 5%. Primary analysis due to result of Shapiro-Wilk test; Test was stratified by region and therapy naive/add-on therapy
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — Additional analysis due to result of Shapiro-Wilk test; Mean Difference (Final Values) = 35.78, 95% CI 2-sided [20.06 to 51.51]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT vs Placebo; Shapiro-Wilk test for normality of ANCOVA residuals; Test type: Superiority or Other; p = 0.0001, Shapiro-Wilk

2. Secondary Outcome: Pulmonary Vascular Resistance (PVR) - Change From Baseline to Week 12
Description: The pulmonary vascular resistance (PVR) is a calculated hemodynamic parameter. PVR is derived from the directly measured parameters mean pulmonary arterial pressure (PAPmean) and pulmonary capillary wedge pressure (PCWP), divided by the cardiac output (CO). PVR and PAPmean are acquired during a right heart catheterization. CO is a calculated hemodynamic parameter, too. Formula: PVR = 80*(PAPmean - PCWP)/CO
Time Frame: Baseline and week 12
Population: Intent to Treat (ITT) - a randomized participant was valid for ITT analyses if at least one dose of study medication was administered. Only participants with a baseline and at least one post-baseline measurement were included in the analysis of PVR.
Measure: Mean (Standard Deviation); unit: dyn*s*cm^-5
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Riociguat (Adempas, BAY63-2521) up to 1.5 mg_IDT | Placebo
Number analyzed (Participants) | 232 | 58 | 107
dyn*s*cm^-5 | -223.29 (260.09) | -167.79 (320.22) | -8.89 (316.57)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT vs Placebo; Missing values at week 12 were imputed using the last available post-baseline observation. Same analysis method as for primary efficacy parameter; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Hierarchical testing for secondary efficacy parameters in the order: PVR, NT-proBNP, WHO functional class, TTCW, Borg scale, EQ5D, LPH. Primary analysis due to result of Shapiro-Wilk test; Test was stratified by region and therapy naive/add-on therapy
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — Additional analysis due to result of Shapiro-Wilk test; Mean Difference (Final Values) = -225.72, 95% CI 2-sided [-281.37 to -170.08]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT vs Placebo; Shapiro-Wilk test for normality of ANCOVA residuals; Test type: Superiority or Other; p = 0.0001, Shapiro-Wilk

3. Secondary Outcome: N-terminal Prohormone of Brain Natriuretic Peptide (NT-proBNP) - Change From Baseline to Week 12
Description: N-terminal pro-brain natriuretic peptide (NT-proBNP) levels in the blood are used for screening, diagnosis of acute congestive heart failure (CHF) and may be useful to establish prognosis in heart failure.
Time Frame: Baseline and week 12
Population: Intent to Treat (ITT) - a randomized participant was valid for ITT analyses if at least one dose of study medication was administered. Only participants with a baseline and at least one post-baseline measurement were included in the analysis of NT-proBNP.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Riociguat (Adempas, BAY63-2521) up to 1.5 mg_IDT | Placebo
Number analyzed (Participants) | 228 | 54 | 106
pg/mL | -197.89 (1721.29) | -471.50 (913.02) | 232.39 (1011.09)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — Hierarchical testing for secondary efficacy parameters in the order: PVR, NT-proBNP, WHO functional class, Time to clinical worsening, Borg scale, EQ5D, LPH. Primary analysis due to result of Shapiro-Wilk test; Test was stratified by region and therapy naive/add-on therapy
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT vs Placebo; Test type: Superiority or Other; p = 0.0157, ANCOVA — Additional analysis due to result of Shapiro-Wilk test; Mean Difference (Final Values) = -431.81, 95% CI 2-sided [-781.52 to -82.10]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT vs Placebo; Shapiro-Wilk test for normality of ANCOVA residuals; Test type: Superiority or Other; p = 0.0001, Shapiro-Wilk

4. Secondary Outcome: World Health Organization (WHO) Functional Class - Change From Baseline to Week 12
Description: The WHO functional assessment of pulmonary arterial hypertension ranged from functional class I (participants with PH but without resulting limitation of physical activity) to class IV (participants with PH with inability to carry out any physical activity without symptoms. These participants manifest signs of right-heart failure.). Changes to a lower WHO functional class resemble improvement; changes to a higher functional class resemble deterioration of PAH.
Time Frame: Baseline and week 12
Population: Intent to Treat (ITT) - a randomized participant was valid for ITT analyses if at least one dose of study medication was administered. Participants with a missing baseline were excluded from the analysis of WHO functional class.
Measure: Number; unit: Percentage of participants
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Riociguat (Adempas, BAY63-2521) up to 1.5 mg_IDT | Placebo
Number analyzed (Participants) | 254 | 63 | 125
Percentage of participants
  -2 | 0.4 | 0 | 0
  -1 | 20.5 | 23.8 | 14.4
  0 | 75.6 | 68.3 | 71.2
  1 | 2.8 | 6.3 | 12.0
  2 | 0.4 | 1.6 | 2.4
  3 | 0.4 | 0 | 0
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT vs Placebo; Missing values for participants who withdrew or died before 12 weeks were imputed with a worst value of IV in case of clinical worsening without termination visit or measurement at that termination visit and with a worst value of V in case of death and with the last observed value otherwise; Test type: Superiority or Other; p = 0.0033, Wilcoxon (Mann-Whitney) — Hierarchical testing for secondary efficacy parameters in the order: PVR, NT-proBNP, WHO functional class, Time to clinical worsening, Borg scale, EQ5D, LPH; Test was stratified by region and therapy naive/add-on therapy

5. Secondary Outcome: Percentage of Participants With Clinical Worsening
Description: The combined endpoint "time to clinical worsening", made up of the following components, defined by the first occurrence: all-cause mortality; heart/lung transplantation; atrial septostomy; first hospitalization due to pulmonary hypertension; start of a new pulmonary hypertension treatment; persistent worsening of 6MWD or WHO functional class due to deterioration of PH .
Time Frame: At week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Riociguat (Adempas, BAY63-2521) up to 1.5 mg_IDT | Placebo
Number analyzed (Participants) | 254 | 63 | 126
Percentage of participants
  Any event | 1.2 | 3.2 | 6.3
  Hospitalization due to pulmonary hypertension | 0.4 | 0 | 3.2
  Start of new pulmonary hypertension treatment | 0.4 | 1.6 | 4.0
  Decrease in 6MWT due to pulmonary hypertension | 0.4 | 1.6 | 1.6
  Persistant worsening of functional class due to PH | 0 | 0 | 0.8
  Death | 0.8 | 1.6 | 2.4
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT vs Placebo; The test is for difference of occurence of "Any event"; Test type: Superiority or Other; p = 0.0046, Log Rank — [p-value comment as in outcome 4, analysis 1]; Test was stratified by region and therapy naive/add-on therapy; Risk Difference (RD) = -5.20, 95% CI 2-sided [-9.85 to -0.55] — Based on Mantel-Haenszel estimate stratified by region and therapy naive/add-on therapy

6. Secondary Outcome: Borg CR 10 Scale - Change From Baseline to Week 12
Description: The Borg CR10 Scale is a participant reported outcome measure used in clinical diagnosis of e.g. breathlessness and dyspnea. It documents the participant's exertion during a physical test. Low values indicate low levels of exertion; high values indicate more intense exertion reported by the participant. The score ranges from 0 ("Nothing at all") to 10 ("Extremely strong - Maximal").
Time Frame: Baseline and week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Riociguat (Adempas, BAY63-2521) up to 1.5 mg_IDT | Placebo
Number analyzed (Participants) | 254 | 63 | 126
Scores on a scale | -0.44 (1.72) | -0.33 (1.47) | 0.09 (2.05)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT vs Placebo; Missing values for participants who withdrew or died before 12 weeks were imputed with a worst value of 10 in case of death or clinical worsening without termination visit and with the last observed value otherwise; Test type: Superiority or Other; p = 0.0022, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 4, analysis 1]; Test was stratified by region and therapy naive/add-on therapy

7. Secondary Outcome: EQ-5D Utility Score - Change From Baseline to Week 12
Description: EQ-5D utility score is a Quality-of-Life participant reported outcome measure. The utility score is calculated based on five questions concerning problems with mobility, self-care, usual activities, pain/discomfort and anxiety/depression. An increase in the utility score represents an improvement in quality of life. The score ranges from -0.594 (worst answer in all five questions) to 1 (best answer in all five questions).
Time Frame: Baseline and week 12
Population: Intent to Treat (ITT) - a randomized participant was valid for ITT analyses if at least one dose of study medication was administered. Participants with a missing baseline were excluded from the analysis of the EQ5D utility score.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Riociguat (Adempas, BAY63-2521) up to 1.5 mg_IDT | Placebo
Number analyzed (Participants) | 253 | 62 | 124
Scores on a scale | 0.0329 (0.2350) | 0.0782 (0.3111) | -0.0317 (0.3044)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT vs Placebo; Missing values at baseline were imputed using last available observation prior to start of study treatment. Missing values for participants who withdrew or died before 12 weeks were imputed with a worst value of -0.594 in case of death or clinical worsening without termination visit and with the last observed value otherwise; Test type: Superiority or Other; p = 0.0663, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 3, analysis 1]; Test was stratified by region and therapy naive/add-on therapy
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT vs Placebo; Test type: Superiority or Other; p = 0.0197, ANCOVA — Additional analysis due to result of Shapiro-Wilk test; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [0.01 to 0.11]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT vs Placebo; Shapiro-Wilk test for normality of ANCOVA residuals; Test type: Superiority or Other; p = 0.0001, Shapiro-Wilk

8. Secondary Outcome: Living With Pulmonary Hypertension (LPH) Questionnaire - Change From Baseline to Week 12
Description: The self-reported Living with Pulmonary Hypertension (LPH) questionnaire is designed to measure the effects of PH and PH-specific treatments on an individual's quality of life. The LPH total score can range from 0 (best) to 105 (worst).
Time Frame: Baseline and week 12
Population: Intent to Treat (ITT) - a randomized participant was valid for ITT analyses if at least one dose of study medication was administered. Participants with a missing baseline were excluded from the analysis of the LPH questionnaire.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Riociguat (Adempas, BAY63-2521) up to 1.5 mg_IDT | Placebo
Number analyzed (Participants) | 247 | 62 | 122
Scores on a scale | -5.99 (17.76) | -10.21 (21.27) | 0.36 (18.15)
Statistical Analysis 1: Comparison: Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT vs Placebo; Missing values at baseline were imputed using last available observation prior to start of study treatment. Missing values for participants who withdrew or died before 12 weeks were imputed with a worst value of 105 in case of death or clinical worsening without termination visit and with the last observed value otherwise; Test type: Superiority or Other; p = 0.0019, Wilcoxon (Mann-Whitney) — Hierarchical testing for secondary efficacy parameters in the order: PVR, NT-proBNP, WHO FC, TTCW, Borg scale, EQ5D, LPH. Primary analysis due to result of Shapiro-Wilk test. Nominally significant only due to hierarchical testing; Test was stratified by region and therapy naive/add-on therapy
Statistical Analysis 2: Comparison: Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT vs Placebo; Test type: Superiority or Other; p = 0.0009, ANCOVA — Additional analysis due to result of Shapiro-Wilk test; Mean Difference (Final Values) = -6.17, 95% CI 2-sided [-9.79 to -2.54]
Statistical Analysis 3: Comparison: Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT vs Placebo; Shapiro-Wilk test for normality of ANCOVA residuals; Test type: Superiority or Other; p = 0.0001, Shapiro-Wilk

ADVERSE EVENTS:
Time Frame: Adverse event data were collected after signing the informed consent until 2 days after end of study treatment over a period of approximately 30 days.
Arm/Group | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT | Riociguat (Adempas, BAY63-2521) up to 1.5 mg_IDT | Placebo
Serious Adverse Events (participants affected / at risk) | 29/254 | 11/63 | 23/126
Other Adverse Events (participants affected / at risk) | 216/254 | 57/63 | 96/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT (N=254) | Riociguat (Adempas, BAY63-2521) up to 1.5 mg_IDT (N=63) | Placebo (N=126)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 2 | 3 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Retinal artery occlusion (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 1
Chest pain (General disorders) | 2 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 1
Encephalitis herpes (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Mycoplasma infection (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Catheterisation cardiac (Investigations) | 1 | 0 | 0
Electrocardiogram ST-T segment abnormal (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 3 | 0 | 5
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Circulatory collapse (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Riociguat (Adempas, BAY63-2521) up to 2.5 mg_IDT (N=254) | Riociguat (Adempas, BAY63-2521) up to 1.5 mg_IDT (N=63) | Placebo (N=126)
Anaemia (Blood and lymphatic system disorders) | 20 | 1 | 3
Palpitations (Cardiac disorders) | 20 | 5 | 6
Tachycardia (Cardiac disorders) | 9 | 0 | 7
Abdominal discomfort (Gastrointestinal disorders) | 7 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 6 | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 9 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 9 | 2 | 5
Constipation (Gastrointestinal disorders) | 9 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 35 | 6 | 12
Dyspepsia (Gastrointestinal disorders) | 48 | 8 | 10
Gastric polyps (Gastrointestinal disorders) | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 3 | 4 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 14 | 4 | 4
Nausea (Gastrointestinal disorders) | 40 | 10 | 16
Vomiting (Gastrointestinal disorders) | 26 | 7 | 11
Asthenia (General disorders) | 6 | 2 | 2
Chest discomfort (General disorders) | 6 | 4 | 11
Chest pain (General disorders) | 16 | 4 | 10
Face oedema (General disorders) | 5 | 1 | 4
Fatigue (General disorders) | 7 | 0 | 8
Feeling hot (General disorders) | 2 | 0 | 3
Oedema (General disorders) | 8 | 1 | 2
Oedema peripheral (General disorders) | 44 | 14 | 14
Pyrexia (General disorders) | 7 | 6 | 4
Bronchitis (Infections and infestations) | 8 | 3 | 3
Gastroenteritis (Infections and infestations) | 7 | 0 | 1
Nasopharyngitis (Infections and infestations) | 26 | 6 | 14
Oral candidiasis (Infections and infestations) | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 7 | 2 | 5
Urinary tract infection (Infections and infestations) | 3 | 0 | 4
Respiratory tract infection (Infections and infestations) | 7 | 2 | 5
Activated partial thromboplastin time prolonged (Investigations) | 3 | 0 | 3
Haemoglobin decreased (Investigations) | 0 | 3 | 0
International normalised ratio increased (Investigations) | 6 | 0 | 5
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 3 | 6
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 5 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 3 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 0 | 6
Dizziness (Nervous system disorders) | 39 | 15 | 15
Headache (Nervous system disorders) | 69 | 20 | 25
Presyncope (Nervous system disorders) | 4 | 2 | 0
Anxiety (Psychiatric disorders) | 2 | 2 | 2
Insomnia (Psychiatric disorders) | 9 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 3 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 4 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 4 | 3
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 3 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 2 | 2
Flushing (Vascular disorders) | 5 | 2 | 7
Hypotension (Vascular disorders) | 24 | 2 | 3
Hot flush (Vascular disorders) | 1 | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The embargo can be up to 6 months (equal to the 180 days), moreover if it is necessary the embargo period can be prolonged to expiry of priority year.